CLINICAL TRIAL: NCT04653701
Title: A Single Center Experience:Safety and Efficacy of DEB-TACE Performed With a Novel Reflux-control Microcatheter in Patients With Early and Intermediate HCC.
Brief Title: Safety and Efficacy of DEB-TACE Performed With a Novel Reflux-control Microcatheter in Patients With HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Juan José Ciampi Dopazo (Other)
Responsible Party: Sponsor-Investigator, Juan José Ciampi Dopazo, Principal Investigator and Clinical Professor, University Hospital Virgen de las Nieves
Organization: University Hospital Virgen de las Nieves (Other)
Other Study IDs: 5077
Record Dates: First submitted 2020-11-15; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: embolization; chemoembolization; superselective embolization
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with hepatocellular carcinoma treated with TAMDEM® 100 micron and SEQURE® microcatheter: Patients included in this study and with chemoembolization indications will be superselective embolized using TAMDEM® 100 micron preloaded particles (Doxorubicin) and SEQURE® microcatheter combination (SYNERGIC EFFECT). Objective tumoral response and 30 days-complications (Safety) are primary outcomes.
  Interventions: Combination Product: Chemoembolization with preloaded microparticles 100 micron and reflux control microcatheter

INTERVENTIONS:
Combination Product: Chemoembolization with preloaded microparticles 100 micron and reflux control microcatheter — We will perform chemoembolization technique in those patients (during 1 year) with indications for this treatment in relation with guidelines (early and intermediate hepatocellular carcinoma). Specific microcatheter and microparticles will be use (Mentioned above)

SUMMARY:
BACKGROUND:

Hepatocellular carcinoma is the fifth most frequent cancer in the world, with a diagnosis of more than 500,000 new cases per year. It is considered the third leading cause of cancer mortality and presents well-defined risk factors. Liver cirrhosis is the main risk factor for developing HCC, therefore screening programs in cirrhotic patients will allow the early diagnosis of this neoplasia. Despite this, most HCCs are diagnosed at a stage in which the application of curative therapies is no longer possible.

Hepatic transarterial chemoembolization (TACE) belongs to the arterially directed embolization therapies for the treatment of unresectable early-to-advanced hepatocellular carcinoma (HCC). It is the only therapy that has shown to improve survival in intermediate-stage HCC.

Drug-eluting beads (DEB)-TACE has shown to provide slow drug elution, reduced liver and systemic toxicity, increased local drug concentration, and tissue necrosis.

Aside from TACE, other transarterial options include bland embolization, or hepatic artery embolization (HAE), and transarterial radioembolization (TARE). All have an acceptable safety profile, and each has its associated procedural and peri-procedural complications. One potential complication that may occur during all embolization procedures is when the embolic material migrates outside of the desired treatment area, leading to non-target embolization (NTE). In fact, when collateral vessels are embolized, there is a risk that these may be feeders of non-target tissue or organs.

NTE following TACE in particular may lead to a double-layer problem: dangerous components affecting healthy tissue, one ischemic and one related to cytotoxicity from the chemotherapeutic agent, which may have clinical consequences, and potential incomplete treatment of the lesion (due to beads being "deviated" from target).

NTE is highly recognized, but often thought to be uncommon, and although different complications can be caused by it, there may appear to be no evidence of NTE during the intraprocedural imaging.

To avoid the complications due to NTE, apart from the importance of the pre-, intra- and post-procedural imaging, and the thorough study of the anatomical picture, the catheters/microcatheters should also be chosen with reason and care. In particular, selective catheterization should be achieved by placing the microcatheter tip as close as possible to the target, through the specific branch/branches supplying it.

However, even with the microcatheter selectively positioned in the vessel to be embolized, the risk of NTE might not be eliminated, since it could happen as a result of changes in flow dynamics that occur during embolization, particularly when the endpoint is stasis. These changes could result in reflux into non-target territories and, as such, might be better prevented with the use of microcatheters intended to reduce reflux. To this purpose, the use of a dedicated delivery device should be taken into consideration, in order to optimize and save time during the procedure.

Microcatheters are commonly used during most arterial embolization procedures, and as explained above, there is a strong rationale to use a reflux-control microcatheter - like Sequre - for DEB-TACE.

The main expectation is to achieve technical success with Sequre in all patients with a reachable target lesion, with the intent not only to minimize potential damage to surrounding tissue, but also to potentially deliver more treatment embolics, as all the beads are (re)directed towards the target.

The use of small diameter particles (100 micron-TANDEM ® spheres), induces superior tumor necrosis response (Urbano et al., European Journal of Radiology, 2020); with the synergistic effect of being administered through the SEQURE anti-reflux protection system, there is reason to believe that it will be possible to administer maximum doses of doxorubicin, while avoiding the occlusion of non-target arterial segments (SYNERGIC EFFECT).

STUDY PROPOSAL:

We propose a prospective observational study with data collection from a single center (Virgen de las Nieves University Hospital-Granada), for a period that ranges October 2020-December 2021. Here summarized the inclusion criteria and contraindications:

Inclusion criteria

* BCLC B and or some case BCLC A
* Both genders
* Over 18 years.
* Bilirubin less than 3 gr/dl.
* No contraindications to the use of iodinated contrast
* Absence of chronic kidney disease
* ECOG 0-1.
* Absence of encephalopathy.
* Informed consent.

Contraindications

* Advanced liver disease.
* Thrombosis or reversal of portal flow.
* Vascular invasion.
* Extrahepatic spread.
* Contraindication to administration of cytostatics.
* Contraindication to angiographic procedure.

DETAILED DESCRIPTION:
Microcatheters are commonly used during most arterial embolization procedures. SEQURE® (Guerbet, France) is an innovative reflux-control microcatheter for peripheral embolization procedures which relies on flow dynamics as the foundation of its' mechanism of action. It can optimize the delivery of calibrated microspheres of specific sizes.

The device presents as a regular microcatheter with a non-tapered internal lumen for delivery of embolics (typically in suspension with contrast media), and 2 radiopaque markers (placed at a distance of 11 mm) at the tip (distal marker being at 0.5-1 mm from the point of exit).

Near the distal atraumatic tip, between the two markers, it has side slits (approximately 50 µm in width) which allow contrast media to exit radially in addition to the standard fluid flow through the distal tip of the catheter. The contrast media that comes out of the side-holes creates a turbulence in the space surrounding the slits, between microcatheter and vessel, which acts as a fluid barrier in that given portion. This fluid-dynamic barrier redirects the beads that tend to upstream reflux back to their flow-directed trajectory, preventing the beads from migrating in non-target areas, and thus eliminating, or strongly reducing, undesired non-target embolization (NTE).

Moreover, SEQURE® allows for haemodynamic arrangement to be preserved, by favoring and maintaining unaltered the natural blood flow. Under fluoroscopy, the radial flow of contrast media exiting through the side holes in the SEQURE® microcatheter can be seen, giving the physician indication of the vessel flow dynamics.

Lesions were identified and then treated supra-selectively with the microcatheter, with the embolic materials infused in a slow and controlled manner, in order to reduce reflux into non-target branches

HYPOTHESIS:

The use of 100 micron-TANDEM ® spheres will be studied with the synergistic effect of being administered through SEQURE® microcatheter anti-reflux protection system, which may allow the administration of the maximum doses of doxorubicin, avoiding the undesired oclussion of collateral arterial segments (SYNERGIC EFFECT) in a prospective study in patients with hepatocellular carcinoma early-intermediate stage.

PATIENT SELECTION:

Between October 2020 and December 2021, and expected number of 30 patients will be treated. The diagnosis of Hepatocellular carcinoma (HCC) will confirm in accordance with the American Association for the Study of Liver Diseases guidelines and HCC staged according to Barcelona Clinic Liver Cancer (BCLC) system.

DEB-TACE is indicated according to clinical practice guidelines referred above.

TECHNICAL PROCEDURE:

The embolization will be performed using TANDEM ® spheres (each cc of spheres can be loaded with up to 50 mg of doxorubicin. The maximum dose of doxorubicin used per procedure was 150 mg, corresponding to 3 cc of spheres) and SEQURE ® microcatheter in a super-selective tumour´s arterial position avoiding undesired arterial branches. The procedure will consider super-selective when the micro-catheter tip reached the tumour feeding artery. Each cc of microspheres will mix with 7-10 cc of non-ionic contrast medium. Embolization endpoint is considered vascular stasis or 150 mg of Doxorubin administered.

OBJECTIVES AND END-POINTS:

Efficacy:

* Technical success will be defined as a composite outcome measurement: ability to place the microcatheter inside the required vascular segment and qualitative assessment of microspheres deposition in the target tumour.
* Time to Progression (TTP) [Time Frame: 6 months]. Time at which progression is first observed in a tumor assessment according to mRECIST as assessed by CT or MRI.
* Objective Response Rate (ORR) and Disease Control Rate (DCR) [Time Frame: Assessed at 1, 3, and 6 months after first treatment]. ORR is defined as a complete or partial response among the total number of cases and DCR is defined as a complete, partial response or stable disease among the total number of cases , according to mRECIST evaluated by CT or MRI. Time to retreatment included as consequential secondary objective.

Safety:

* Adverse Events (AEs) and Serious Adverse Events (SAE) [Time Frame: Assessed at 1, 3, and 6 months after first treatment. The incidence of emerging AE and SAE will be summarized according to standardized qualification criteria [Journal of Vascular Interventional Radiology (JVIR) SAE], including pancreatitis, cholecystitis, clinical presentations, postembolization syndrome (PES), etc.
* Non Target embolization (NTE) by thorough angiographic assessment of the whole liver vasculature after TACE, as well as Cone Beam Computed Tomography (CBCT) performed immediately following embolization (within 30 minutes from the end of procedure) to evaluate off-target distribution.
* Health-Related Quality of Life questionary (HRQOL): pre-treatment and post-treatment quality of life assessment using the specific questionnaire for functional assessment for cancer treatment (FACT-G).

DATA COLLECTION AND FOLLOW-UP:

The information will be collected through the electronic database of the patient (includes laboratory data). Patients will be evaluated starting from the date of inclusion as candidates for TACE treatment, and followed up for 6 months (unless patients are lost to clinical follow-up or death occurs). Mortality data are obtainable by searching the electronic history of the patient.

Changes in the serum levels of aspartate aminotransferase (AST), alanine aminotransferase (ALT), Alkaline phosphatase (ALP), bilirubin, albumin and patients' complete hematological profile, as well as serum lipase and amylase levels within the 1st week post-TACE to detect pancreatitis, will be evaluated at the following time-points: pre-embolization, at one month, three months, and six months. Computed tomography (CT) or Magnetic Resonance Imaging (MRI) with contrast will be performed at the same time-points as just indicated; modified Response Evaluation Criteria in Solid Tumors ( m-RECIST) will be used, and images will be assessed by two experienced radiologists (any discordant interpretation will be solved through team consensus). All serologic toxicities would be classified according to common terminology criteria for adverse effects. On this scale, severe hepato-toxicity (grade 3) is classified as the increase of up to 5 times the normal limit of AST, ALT, FA or the increase of bilirubin level to over 3 g/dl.

ELIGIBILITY:
Inclusion Criteria:

* BCLC B and or some case BCLC A
* Both genders
* Over 18 years.
* Bilirubin less than 3 gr/dl.
* No contraindications to the use of iodinated contrast
* Absence of chronic kidney disease
* ECOG 0-1.
* Absence of encephalopathy.
* Informed consent.

Exclusion Criteria:

* Advanced liver disease.
* Thrombosis or reversal of portal flow.
* Vascular invasion.
* Extrahepatic spread.
* Contraindication to administration of cytostatics.
* Contraindication to angiographic procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be evaluated starting from the date of inclusion as candidates for TACE treatment, and followed up for 6 months . Mortality data are obtainable by searching the electronic history of the patient.
  Changes in the serum levels of AST, ALT, FA, bilirubin, albumin and patients' complete hematological profile, as well as serum lipase and amylase levels within the 1st week post-TACE to detect pancreatitis, will be evaluated at the following time-points: pre-embolization, at one month, three months, and six months. CT or MRI with contrast will be performed at the same time-points as just indicated; m-RECIST criteria will be used. All serologic toxicities would be classified according to common terminology criteria for adverse effects.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-11-14 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2022-02-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Assessed at 3 months after patient inclusion
  ORR is defined as a complete or partial response among total of treated cases, according to mRECIST evaluated by CT or MRI. The value of these data is a percentage considering tumour diameter before and after treatment.
Objective Response Rate (ORR) | Assessed at 6 months after patient inclusion
  ORR is defined as a complete or partial response among total of treated cases, according to mRECIST evaluated by CT or MRI. The value of these data is a percentage considering tumour diameter before and after treatment.
Disease Control Rate (DCR) | Assessed at 3 months after patient inclusion
  DCR is defined as a complete, partial response or stable disease among total of treated cases, according to mRECIST evaluated by CT or MRI. The value of these data is a percentage considering tumour diameter before and after treatment.
Disease Control Rate (DCR) | Assessed at 6 months after patient inclusion
  DCR is defined as a complete, partial response or stable disease among total of treated cases, according to mRECIST evaluated by CT or MRI. The value of these data is a percentage considering tumour diameter before and after treatment.
Adverse Events (AEs) and Serious Adverse Events (SAE) | Assessed up to 30 days after patient inclusion
  The incidence of emerging AE and SAE will be summarized according to standardized qualification criteria (JVIR SAE), including pancreatitis, cholecystitis, clinical presentations, PES, etc.
Technical success | up to 1 hour after patient inclusion (or after patient treatment)
  Defined as a composite outcome measurement: ability to place the micro-catheter inside the required vascular segment and qualitative assessment of microspheres deposition in the target tumour.

CONTACTS AND LOCATIONS:
Overall Officials: JUAN JOSE CIAMPI DOPAZO, Dr, Principal Investigator — University Hospital Virgen de las Nieves
Locations (1):
- Juan Jose Ciampi Dopazo, Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Between September 2021 to March 2022

REFERENCES:
- [Background] Delicque J, Guiu B, Boulin M, Schwanz H, Piron L, Cassinotto C. Liver chemoembolization of hepatocellular carcinoma using TANDEM(R) microspheres. Future Oncol. 2018 Nov;14(26):2761-2772. doi: 10.2217/fon-2018-0237. Epub 2018 Jun 28. PMID 29953255
- [Result] Lammer J, Malagari K, Vogl T, Pilleul F, Denys A, Watkinson A, Pitton M, Sergent G, Pfammatter T, Terraz S, Benhamou Y, Avajon Y, Gruenberger T, Pomoni M, Langenberger H, Schuchmann M, Dumortier J, Mueller C, Chevallier P, Lencioni R; PRECISION V Investigators. Prospective randomized study of doxorubicin-eluting-bead embolization in the treatment of hepatocellular carcinoma: results of the PRECISION V study. Cardiovasc Intervent Radiol. 2010 Feb;33(1):41-52. doi: 10.1007/s00270-009-9711-7. Epub 2009 Nov 12. PMID 19908093
- [Result] Urbano J, Echevarria-Uraga JJ, Ciampi-Dopazo JJ, Sanchez-Corral JA, Cobos Alonso J, Anton-Ladislao A, Pena-Baranda B, Nacarino-Mejias V, Gonzalez-Costero R, Munoz Ruiz-Canela JJ, Perez-Cuesta J, Lanciego C, de Gregorio MA. Multicentre prospective study of drug-eluting bead chemoembolisation safety using tightly calibrated small microspheres in non-resectable hepatocellular carcinoma. Eur J Radiol. 2020 May;126:108966. doi: 10.1016/j.ejrad.2020.108966. Epub 2020 Mar 19. PMID 32278280
- [Result] Aliberti C, Carandina R, Lonardi S, Dadduzio V, Vitale A, Gringeri E, Zanus G, Cillo U. Transarterial Chemoembolization with Small Drug-Eluting Beads in Patients with Hepatocellular Carcinoma: Experience from a Cohort of 421 Patients at an Italian Center. J Vasc Interv Radiol. 2017 Nov;28(11):1495-1502. doi: 10.1016/j.jvir.2017.07.020. Epub 2017 Sep 18. PMID 28927662
- [Result] Lopez-Benitez R, Richter GM, Kauczor HU, Stampfl S, Kladeck J, Radeleff BA, Neukamm M, Hallscheidt PJ. Analysis of nontarget embolization mechanisms during embolization and chemoembolization procedures. Cardiovasc Intervent Radiol. 2009 Jul;32(4):615-22. doi: 10.1007/s00270-009-9568-9. Epub 2009 Apr 23. PMID 19387732

DOCUMENTS (1):
  • Study Protocol (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT04653701/Prot_000.pdf